CLINICAL TRIAL: NCT02352883
Title: Prospective Study of Magnetic Resonance Imaging (MRI) and Multiparameter Gene Expression Assay in Ductal Carcinoma In Situ (DCIS)
Brief Title: MRI and Gene Expression in Diagnosing Patients With Ductal Breast Cancer In Situ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: E4112; NCI-2014-01261 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E4112 (Other: ECOG-ACRIN Cancer Research Group); ECOG-E4112 (Other: DCP); UG1CA189828 (NIH); U10CA037403 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-02-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ductal Breast Carcinoma In Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Steroids

ARMS (5):
- Arm A (MRI) (Experimental): Patients undergo MRI prior to surgery. Patients undergo additional imaging and/or biopsies if indicated based on MRI.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis; Other: Cytology Specimen Collection Procedure
- Arm B (mastectomy) (Experimental): Patients undergo a mastectomy. Patients do not register for Step 3.
  Interventions: Procedure: Therapeutic Conventional Surgery; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis; Other: Cytology Specimen Collection Procedure
- Arm C (wide local excision) (Experimental): Patients undergo wide local excision +/- re-excision. Patients may cross-over to Arm B if mastectomy is indicated. Tissue samples collected during surgery are used to calculate the DCIS score using genetic analysis testing. Patients may then proceed to Step 3.
  Interventions: Procedure: Therapeutic Surgical Procedure; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis; Other: Cytology Specimen Collection Procedure
- Arm D (endocrine therapy) (Experimental): Patients undergo endocrine therapy as directed.
  Interventions: Drug: Endocrine Therapy; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis; Other: Cytology Specimen Collection Procedure
- Arm E (radiation therapy, endocrine therapy) (Experimental): Patients undergo radiation therapy and endocrine therapy as directed.
  Interventions: Radiation: Radiation Therapy; Drug: Endocrine Therapy; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; MRI; MRI Scan; NMRI
  Arms: Arm A (MRI)
Procedure: Therapeutic Conventional Surgery — Undergo mastectomy
  Arms: Arm B (mastectomy)
Procedure: Therapeutic Surgical Procedure — Undergo wide local excision
  Arms: Arm C (wide local excision)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT
  Arms: Arm E (radiation therapy, endocrine therapy)
Drug: Endocrine Therapy — Undergo endocrine therapy
  Other Names: Chemotherapy-Hormones/Steroids; Hormonal Therapy; Hormone Therapy
  Arms: Arm D (endocrine therapy); Arm E (radiation therapy, endocrine therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
  Arms: Arm A (MRI); Arm B (mastectomy); Arm C (wide local excision); Arm D (endocrine therapy)

SUMMARY:
This clinical trial studies magnetic resonance imaging (MRI) and gene expression in diagnosing patients with abnormal cells in the breast duct that have not spread outside the duct. MRI uses radio waves and a powerful magnet linked to a computer to create detailed pictures of areas inside the body. MRI may help find and diagnose patients with breast cancer. It may also help doctors predict a patient's response to treatment and help plan the best treatment. Genetic studies may help doctors predict the outcome of treatment and the risk for disease recurrence. Performing MRI with genetic studies may help determine the best treatment for patients with breast cancer in situ.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with ductal carcinoma in situ (DCIS) diagnosed on core needle biopsy judged to be breast conservation candidates based upon standard imaging (mammography +/- sonography) and physical examination (a) who convert to mastectomy in step 1 based on MRI findings, and (b) who have a mastectomy as the final surgical procedure in step 2.

SECONDARY OBJECTIVES:

I. To assess the relation between baseline clinical covariates (e.g., tumor grade, necrosis, histologic type, mammographic lesion size), MRI morphologic and kinetic features, and the DCIS score.

II. To assess the diagnostic accuracy of MRI in extent of disease evaluation in patients with DCIS.

III. To estimate the proportion of patients who require re-operation because of inadequate excision after MRI.

IV. To estimate the proportion of patients who proceed to mastectomy after an initial attempt at wide local excision because of either inadequate tumor-free margins (< 2 mm), or other reasons.

V. To estimate the 5-year and 10-year ipsilateral breast event (in situ and invasive) rate (IBE) among women with DCIS assessed with MRI preoperatively and treated with wide local excision without radiation therapy (if there is a low DCIS score) or with radiation therapy (if there is an intermediate-high DCIS score).

VI. To estimate the proportion of women with DCIS who receive treatment that is concordant with their treatment goals and concerns.

VII. To estimate the proportion of women with DCIS whose decision autonomy preference was concordant with perceived level of decision involvement.

VIII. To assess decision quality using knowledge score and decision process. IX. To assess concordance between decision autonomy preference and perceived level of decision involvement, knowledge and decision process scores as independent predictors of decision satisfaction at the first post-operative visit.

X. To assess the relationship of patient-reported outcomes and disease-specific covariates, and quality of life after treatment.

XI. To assess the role of disease status, diagnostic test results and surgeon recommendation as predictors of treatment received.

XII. To compare the patient-reported diagnostic testing burden of bilateral mammography and MRI as measured by Testing Morbidities Index (TMI).

OUTLINE:

STEP 1:

ARM A: Patients undergo MRI prior to surgery. Patients undergo additional imaging and/or biopsies if indicated based on MRI.

STEP 2: Patients are assigned to 1 of 2 treatment arms based on the results of the MRI.

ARM B: Patients undergo a mastectomy. Patients do not register for Step 3.

ARM C: Patients undergo wide local excision +/- re-excision. Patients may cross-over to Arm B if mastectomy is indicated. Tissue samples collected during surgery are used to calculate the DCIS score using genetic analysis testing. Patients may then proceed to Step 3.

STEP 3: Patients are assigned to 1 of 2 treatment arms based on the results of the DCIS score test.

ARM D (DCIS score < 39): Patients undergo endocrine therapy as directed.

ARM E (DCIS score >= 39): Patients undergo radiation therapy and endocrine therapy as directed.

After completion of study treatment, patients are followed up every 6 months for 5 years and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Registration to Step 1:
* Patients must have pathologically confirmed diagnosis of unilateral ductal carcinoma in situ with no evidence of microinvasive or invasive disease obtained by core needle biopsy within 4 months of registration; patients diagnosed by surgical excision are not eligible; patients with synchronous bilateral disease are not eligible; patients with synchronous bilateral disease (i.e., synchronous DCIS or invasive cancer) are not eligible

  * Patients will be staged prior to registration according to the clinical staging criteria adapted from the American Joint Committee on Cancer (AJCC) Cancer Staging Data Forms of the AJCC Cancer Staging Manual, 7th Edition, 2009; Note: For consistency purposes, AJCC 7th Edition will continue to be used throughout the entire study enrollment period
* Required studies include a bilateral screening mammogram within 6 months and diagnostic mammogram of the affected breast within 3 months prior to registration
* Patients must not have previous ipsilateral invasive breast cancer or DCIS
* Patients must not have known deleterious mutations in breast cancer (BRCA) genes
* Patients must not have received hormonal therapy (i.e., tamoxifen, raloxifene, and/or aromatase inhibitors) for prevention of breast cancer within 3 months of the biopsy documenting DCIS
* Patients must not have history of chemotherapy for cancer within 6 months prior to registration
* No prior history of breast radiotherapy that will prevent the use of radiotherapy for the present DCIS
* Patients must be judged to be suitable to undergo MRI and receive the contrast agent gadolinium (exclusions follow):

  * No history of untreatable claustrophobia;
  * No presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants);
  * No history of sickle cell disease;
  * No contraindication to intravenous contrast administration;
  * No known allergy-like reaction to gadolinium or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR); patient may be eligible if willing to undergo pre-treatment as defined by the institution's policy and/or ACR guidance;
  * No findings consistent with renal failure, as determined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m^2 based on a serum creatinine level obtained within 28 days prior to registration;
  * Weight lower than that allowable by the MRI table;
* No prior MRI of the breasts within the 6 months prior to registration
* Patients must be eligible for breast-conserving therapy (BCT) based on clinical examination and mammography; if ultrasound is performed, findings must also be consistent with eligibility for BCT
* Patients must not have multicentric disease scheduled to undergo multiple lumpectomies; multifocal disease that can be encompassed in a single operative bed are eligible
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 3 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study
* Registration to Step 2:
* MRI has been performed in Step 1, and additional imaging studies and biopsies performed if indicated
* The clinician/patient has made the decision as to whether the patient will proceed to wide local excision or mastectomy
* Registration to Step 3:
* Patient's most recent surgery was wide local excision with or without re-excision and for which there was obtained clear (>= 2 mm) margins at breast conserving surgery, and the pathology reveals pure DCIS; patients with invasive cancer or DCIS with microinvasion will not be registered on step 3, but will be followed for clinical outcomes
* The OncotypeDX Patient Report of the DCIS Score from the OncotypeDX Breast Cancer Assay performed by Genomic Health on the excision tissue have been uploaded by the site into the Rave electronic case report forms (eCRF)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients judged to be breast conservation candidates based upon standard imaging and physical examination who convert to mastectomy in step 1 based on MRI findings | After MRI (within 30 days following study entry), and prior to surgery
Proportion of patients judged to be breast conservation candidates based upon standard imaging and physical examination who have a mastectomy as the final surgical procedure in step 2 | Up to 12 months post-op

SECONDARY OUTCOMES:
Factors associated with DCIS score | After surgery (DCIS Score is determined from surgical specimen)
  The relation between baseline clinical covariates (tumor grade, necrosis, histologic type, mammographic lesion size), MRI morphologic and kinetic features, and the DCIS score will be assessed.
Diagnostic accuracy of MRI in extent of disease evaluation in patients with DCIS | Up to 12 months post-op
Proportion of patients who require re-operation because of inadequate excision after MRI | Up to 12 months post-op
  A two-sided 95% Wilson confidence interval will be derived.
Proportion of patients who proceed to mastectomy after an initial attempt at wide local excision because of either inadequate tumor-free margins (< 2mm), or other reasons | Up to 12 months post-op
  A two-sided 95% Wilson confidence interval will be derived. In addition to the overall probability of conversion in this cohort, estimates will be stratified by the reason for conversion.
IBE rate | At 5 years
  Kaplan-Meier curves will be derived for the time to ipsilateral breast event for patients assigned to be treated with RT and those not treated with RT. Point estimates and 95% two-sided confidence intervals will be developed.
IBE rate | At 10 years
  Kaplan-Meier curves will be derived for the time to ipsilateral breast event for patients assigned to be treated with RT and those not treated with RT. Point estimates and 95% two-sided confidence intervals will be developed.
Proportion of women who receive treatment that is concordant with their treatment goals and concerns | Up to 24 months post-op
  The proportion of patients with concordant care will be calculated and a 95% Wilson confidence interval will also be derived.
Proportion of women whose decision autonomy preference was concordant with perceived level of decision involvement | Up to 5 days after pre-surgical consultation
  Concordance will be defined as an exact match between decision autonomy preference (patient-based, shared, surgeon-based) and perceived level of decision involvement (patient based, shared, surgeon-based) as assessed by the Control Preferences Scale, reduced to three categories. The proportion of patients with concordance will be calculated for the sample. In addition, the degree of concordance over the group will be determined using kappa analysis.
Decision quality, assessed using the composite of knowledge score and decision process score | Up to 5 days after pre-surgical consultation
  To calculate knowledge score, a point for each correct answer on the knowledge questionnaire will be assigned, with missing responses receiving 0 points. A total score will be calculated for all patients who complete at least half of the items and scaled from 0-100%. To calculate a decision process score, a point will be assigned for each "yes" or "a lot/some" response. The sum will be scaled from 0-100%. The average of the two scores will be used as the outcome measure.
Role of concordance between decision autonomy preference and perceived level of decision involvement, knowledge and decision process scores as independent predictors of decision satisfaction | Assessed via questionnaire administered at first post-operative visit
  Linear regression modeling will be used in which the response variable will be decision satisfaction. The independent variables will be the indicator of concordance between decision autonomy preference and perceived level of decision involvement, the knowledge score and the decision process score. Two-way interactions between predictors will also be examined.
Patient-reported quality of life, measured using the Patient Reported Outcomes Measurement Information System (PROMIS)10 instrument | At 12 months post-op
  The relationship of patient-reported outcomes and disease specific covariates, and quality of life will be assessed.
Patient-reported quality of life, measured using the PROMIS10 instrument | At 24 months post-op
  The relationship of patient-reported outcomes and disease specific covariates, and quality of life will be assessed.
Role of disease status, diagnostic test results, and surgeon recommendation as predictors of treatment received | Up to 24 months post-op
  Logistic regression modeling will be used in which the response variable will be the indicator of conversion to mastectomy (vs lumpectomy). The independent variables will include covariates describing disease status at baseline, MRI results, surgeon recommendation, patient decision involvement (such as the decision autonomy preference scale) and treatment concerns (as measured via the 7-item questionnaire). Separate analyses will be performed for conversion to mastectomy directly post MRI and conversion to mastectomy following BCS as the response variable.
Patient-reported diagnostic testing burden of bilateral mammogram, MRI, and biopsies, measured by TMI | Up to 5 days after pre-surgical consultation
  A Wilcoxon signed rank test will be used to compare TMI scores for mammography and MRI. In a secondary analysis regression modeling will be used to examine the effects of patient characteristics on the patient's perception of diagnostic test burden for the two modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Lehman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (76):
- United States (76):
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Greenwich Hospital, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Northwestern University, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - IU Health West Hospital, Avon, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Aultman Health Foundation, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

REFERENCES:
- [Derived] Khan SA, Romanoff J, Gatsonis C, Rahbar H, Carlos R, Badve S, Wright J, Corsetti RL, Lehman CD, Spell DW, Han LK, Bumberry JR, Gareen I, Snyder BS, Wagner LI, Miller KD, Comstock C, Sparano JA. Radiotherapy With a 12-Gene Expression Assay for Ductal Carcinoma In Situ: A Randomized Clinical Trial. JAMA Oncol. 2025 Dec 1;11(12):1507-1511. doi: 10.1001/jamaoncol.2025.4079. PMID 41100122
- [Derived] Dunsmore VJ, Snyder BS, Gareen IF, Lehman CD, Khan SA, Romanoff J, Gatsonis C, Corsetti RL, Rahbar H, Spell DW, Han LK, Bumberry JR, Miller KD, Sparano JA, Comstock C, Park E, Wagner LI, Carlos RC. Quality of Life Among Patients With Ductal Carcinoma In Situ. JAMA Netw Open. 2025 Jul 1;8(7):e2518887. doi: 10.1001/jamanetworkopen.2025.18887. PMID 40608342
- [Derived] Slavkova KP, Kang R, Kazerouni AS, Biswas D, Belenky V, Chitalia R, Horng H, Hirano M, Xiao J, Corsetti RL, Javid SH, Spell DW, Wolff AC, Sparano JA, Khan SA, Comstock CE, Romanoff J, Gatsonis C, Lehman CD, Partridge SC, Steingrimsson J, Kontos D, Rahbar H. MRI-based Radiomic Features for Risk Stratification of Ductal Carcinoma in Situ in a Multicenter Setting (ECOG-ACRIN E4112 Trial). Radiology. 2025 Apr;315(1):e241628. doi: 10.1148/radiol.241628. PMID 40167440
- [Derived] Lehman CD, Gatsonis C, Romanoff J, Khan SA, Carlos R, Solin LJ, Badve S, McCaskill-Stevens W, Corsetti RL, Rahbar H, Spell DW, Blankstein KB, Han LK, Sabol JL, Bumberry JR, Gareen I, Snyder BS, Wagner LI, Miller KD, Sparano JA, Comstock C. Association of Magnetic Resonance Imaging and a 12-Gene Expression Assay With Breast Ductal Carcinoma In Situ Treatment. JAMA Oncol. 2019 Jul 1;5(7):1036-1042. doi: 10.1001/jamaoncol.2018.6269. PMID 30653209